CLINICAL TRIAL: NCT03340116
Title: Measurement of Plasma Volume, RBC Volume, and Total Blood Volume Using Daxor Blood Volume Analyzer (BVA-100) in Burn Surgery Patients Pre-operatively and Post-operatively to Determine if Blood Loss During Burn Surgery is Primarily Due to Either Loss of RBC Volume or Hemodilution
Brief Title: Measurement of Blood Volume Loss During Burn Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Unable to find any suitable patients to enroll
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Daxor Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: HM20015231; HM20011159 (Other: VCU IRB)
Record Dates: First submitted 2017-11-01; First posted 2017-11-13 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Surgical Blood Loss; Burns
MeSH Terms: conditions — Blood Loss, Surgical; Burns | interventions — Plasma Volume

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples drawn via venipuncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Pre-operative cohort: This cohort will have their total blood volume, RBC volume, and plasma volumes measured using the Daxor BVA-100 prior to any surgical intervention
  Interventions: Diagnostic Test: Measurement of RBC volume, plasma volume, and total blood volume using Daxor BVA-100
- Post-operative cohort: This cohort will consist of the same study participants in the pre-operative cohort. The only difference is that this cohort will have their total blood volume, RBC volume, and plasma volumes measured using the Daxor BVA-100 AFTER burn surgery.
  Interventions: Procedure: Burn surgery; Diagnostic Test: Measurement of RBC volume, plasma volume, and total blood volume using Daxor BVA-100

INTERVENTIONS:
Procedure: Burn surgery — Burn surgery including wound debridement, skin grafting
  Groups: Post-operative cohort
Diagnostic Test: Measurement of RBC volume, plasma volume, and total blood volume using Daxor BVA-100 — Measurement of RBC volume, plasma volume, and total blood volume using Daxor BVA-100

SUMMARY:
Burn surgery is associated with significant reductions in hematocrit. However, it is unclear whether these reductions are the result of hemodilution from non-red cell containing intraoperative transfusions or from loss of red blood cells. The investigators will be using the Daxor Blood Volume Analyzer (BVA-100), an FDA approved instrument that can measure total blood volume, plasma volume, and RBC volume using the indicator dilution technique. By comparing pre-operative measurements of blood volume, plasma volume, and RBC volume to that of post-operative measurements after burn surgery, the investigators can determine the primary cause of the reduction in hematocrit associated with burn surgery. The investigators hypothesize that these reductions in hematocrit are primarily the result of hemodilution rather than blood loss and that there will be a statistically significant difference in measured plasma volume from the pre-operative group to the post-operative group.

DETAILED DESCRIPTION:
Burn surgery is associated with significant changes (reductions) in hematocrit. However, it is unclear whether these reductions are the result of hemodilution from non-red cell containing intraoperative transfusions or from loss of red blood cells. The investigators will be using the Daxor Blood Volume Analyzer (BVA-100), an FDA approved instrument that can measure total blood volume, plasma volume, and RBC volume using the indicator dilution technique. With this technique, a tracer substance (I-131 albumin) is mixed with an unknown volume. An identical amount of the tracer is mixed into a solution with a known volume. By comparing the concentration of the indicator between the known and unknown volumes, the investigators can determine the volume of the unknown volume (or in this case, the blood volume).

The investigators will be measuring the change in blood volume, plasma volume, and RBC volume from the pre-operative to the post-operative state after completion of burn surgery. We hypothesize that these reductions in hematocrit are primarily the result of hemodilution rather than blood loss and that there will be a statistically significant change in measured plasma volume from the pre-operative to the post-operative measurements.

Average plasma volume for male and female patients is 2950ml SD=590 ml. To detect a 10% increase in plasma volume from hemodilution with a power 0.80 and alpha error 0.05, a one tailed normal distribution t-test determines a sample size fifty. To account for a 10% data loss (technical difficulty, patient withdraw) a sample size of fifty-five would be required.

Fifty-five consecutive adult patients (18 years or older) having burn surgery will be enrolled. Patients with recognized coagulopathy will be excluded. The outcome variables included blood volume (BV, ml), plasma volume (PV, ml) and red blood cell volume (RBCV, ml). All three outcome variables will be measured at two time points; pre-surgery and post-surgery. The pre-surgery measurement will be collected precisely after induction of general anesthesia but prior to surgery start. The post-surgery measurement will be taken immediately after the operation and after all intraoperative red blood cell transfusions are complete. For those patients receiving blood transfusions in the operating room prior to all data collection points, the transfused RBC volume will be recorded and subtracted from the RBCV measured after the transfusion. Transfused RBCV will take into account Hct of 60% for pRBCs. Additional baseline information, including age (year), sex (male, female), weight (kg), and surgery type, will be collected. For the tracer dilution method, the following blood samples will be collected: a baseline (no radiation sample), a first sample 12 minutes after injection (after complete mixing in the blood volume) and additional samples every 6 minutes for at least three successive timed sample points. These multiple timed sample points produce a logarithmic curve of radiation over time, as only a small fraction of albumin leaves the blood volume into the interstitial space. The investigators will compare the pre-operative and post-operative blood volume, RBC volume, and plasma volume measurements to determine if the decrease in hematocrit associated with burn surgery is truly due to hemodilution or loss of RBC volume.

ELIGIBILITY:
Inclusion Criteria:

* Sustained thermal burn of a depth that is deep partial thickness to full thickness and requires operative management
* Burn excision must occur within one week of thermal injury
* Burn size between 10-50% of total body surface area
* Must survive initial resuscitation
* Must consent for blood product transfusion
* Male or non-pregnant female

Exclusion Criteria:

* Cause of burn other than thermal injury (ie electrical or chemical injury)
* Women who are nursing, pregnant, or think they may be pregnant
* Patients with recognized coagulopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18-70 year old male or non-pregnant females who have sustained deep partial thickness to full thickness thermal burns between 10-50% TBSA who are undergoing burn surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change in measured plasma volume | Pre-operative period after intubation, but before surgery start and post-operative period after surgery stop and after all intraoperative blood transfusions are complete
  Measured plasma volume using Daxor BVA-100
Change in measured RBC volume | Pre-operative period after intubation, but before surgery start and post-operative period after surgery stop and after all intraoperative blood transfusions are complete
  Measured RBC volume using Daxor BVA-100
Change in measured total blood volume | Pre-operative period after intubation, but before surgery start and post-operative period after surgery stop and after all intraoperative blood transfusions are complete
  Measured total blood volume using Daxor BVA-100

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nelson, MD, Principal Investigator — VCU Medical Center; Michael Feldman, MD, Principal Investigator — VCU Medical Center

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers outside of the investigators listed in this study group.

REFERENCES:
- [Background] Ong YS, Samuel M, Song C. Meta-analysis of early excision of burns. Burns. 2006 Mar;32(2):145-50. doi: 10.1016/j.burns.2005.09.005. Epub 2006 Jan 18. PMID 16414197
- [Background] Budny PG, Regan PJ, Roberts AH. The estimation of blood loss during burns surgery. Burns. 1993 Apr;19(2):134-7. doi: 10.1016/0305-4179(93)90036-8. PMID 8471147
- [Background] Meiser A, Casagranda O, Skipka G, Laubenthal H. [Quantification of blood loss. How precise is visual estimation and what does its accuracy depend on?]. Anaesthesist. 2001 Jan;50(1):13-20. doi: 10.1007/s001010050957. German. PMID 11220251
- [Background] CRISPELL KR, PORTER B, NIESET RT. Studies of plasma volume using human serum albumin tagged with radioactive iodine. J Clin Invest. 1950 May;29(5):513-6. doi: 10.1172/JCI102288. No abstract available. PMID 15415456
- [Background] Manzone TA, Dam HQ, Soltis D, Sagar VV. Blood volume analysis: a new technique and new clinical interest reinvigorate a classic study. J Nucl Med Technol. 2007 Jun;35(2):55-63; quiz 77, 79. doi: 10.2967/jnmt.106.035972. Epub 2007 May 11. PMID 17496003
- See also: I-131 albumin Volumex Package Insert — http://www.daxor.com/wp-content/uploads/2014/10/volumex-package-insert.pdf